CLINICAL TRIAL: NCT04153071
Title: Evaluation of the Cutaneous Effects of a Unipolar Microplasma Electrode Pin Radiofrequency Device: An In-vivo Histologic Study
Brief Title: Unipolar Microplasma Radiofrequency Device: In-vivo Histologic Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per Investigator and sponsor decision
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALM-OPUS-19-010
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2019-11

CONDITIONS: Skin Resurfacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Unipolar microplasma RF treatment (Experimental): Single cutaneous unipolar microplasma RF treatment, with variable treatment parameters
  Interventions: Device: OPUS system

INTERVENTIONS:
Device: OPUS system — Each subject will have a single cutaneous treatment of their lower abdomen, with variable treatment parameters. Punch biopsies will be obtained from each treatment section, for in-vivo histological evaluations.

SUMMARY:
Prospective, Open-Label, Single-Center Pilot Study.

The study is aimed to evaluate the histologic effects of a unipolar microplasma electrode pin radiofrequency device (Alma Lasers OPUS system) on the abdominal skin.

The study will include up to 2 subjects. Each subject will have a single cutaneous treatment of their lower abdomen, with variable treatment parameters. Punch biopsies will be obtained from each treatment section, for in-vivo histological evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Subject seeking surgical correction of abdominal tissue laxity with an abdominoplasty within the subsequent 1-12 months.
2. Subject abdominal skin must be of appropriate quality to allow for proper study treatment, as judged by the Investigator.
3. The subject must be willing to have punch biopsy specimens obtained from all treated areas following treatment.
4. The Subject must sign a statement of informed consent to the Investigator and Sponsor.

Exclusion Criteria:

1. The subject is less than 18 or greater than 75 years of age.
2. Subject with excessive superficial skin laxity and/or striae of the abdomen, which would prevent proper study treatment.
3. A subject that is unwilling to have punch biopsy specimens obtained from treated areas.
4. Subject with a history of allergy to lidocaine or epinephrine.
5. Known history of keloids or bleeding/coagulation disorder.
6. Presence of surgical or non-surgical scars in the area to be treated.
7. Active inflammatory or infectious process or any other active or serious skin disease in the area to be treated.
8. Planned surgical procedures with incisions and suturing in the area to be treated during the course of the study.
9. Subjects who have had (or plan to have during the course of the study) an abdominal skin treatment with any exclusionary treatments, medications, and/ or devices.
10. Subjects who have used oral isotretinoin or other oral retinoids during the study in the prior 12 months or planning to be on them during the course of the study.
11. Subjects receiving antiplatelet, anticoagulant, or non-steroidal anti-inflammatory agents within 2 weeks of treatment, or planning to receive during the course of the study; in whom, in the Investigator's opinion, administration of radiofrequency treatment may cause procedure-related complications.
12. Women who are pregnant, nursing or intend to become pregnant over the duration of the study, or women who are of childbearing potential not protected by an effective contraceptive method of birth control. Pregnancy status should be checked by urine testing at baseline (Day 0).
13. Subjects who are unwilling or unable to give written consent to participate in the study or unable to comply with the requirements of the clinical trial protocol.
14. Subjects who have received an experimental drug or device within the previous 3 months prior to enrollment.
15. Subjects who are known as alcohol or drug abusers.
16. Subjects who are suffering from any physical or psychological condition, or are under treatment for any such condition which, in the opinion of the Investigator, may constitute an unwarranted risk or which may affect the subjects' compliance or adherence to study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Diameter and depth of ablation and/or coagulation from varying RF device treatment parameters | Immediately post treatment
  Histology analysis to evaluate the diameter and depth of ablation and/or coagulation from varying microplasma RF device treatment parameters, based on biopsy specimens

SECONDARY OUTCOMES:
Rate of adverse events | 10 days
  Safety will be monitored by documentation of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Friedmann, MD, FAAD, Principal Investigator — Westlake Dermatology Clinical Research Center
Locations (1):
- Westlake Dermatology Clinical Research Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No